CLINICAL TRIAL: NCT05061173
Title: Compare the Effects of Aerobic, Resistance, and Combined Training in Overweight/Obese Hypertensive Adults
Brief Title: Comparison of Aerobic, Resistance, and Combined Training in Overweight/Obese Hypertensive Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REC/01083 Sidra Asghar
Record Dates: First submitted 2021-09-18; First posted 2021-09-29 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Obese; Hypertension
Keywords: Aerobic Exercise; Resistive exercise; Combined Aerobic and Resistive Exercise
MeSH Terms: conditions — Obesity; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic exercise training Group (Experimental)
  Interventions: Other: Aerobic exercise training Group
- Resistance Exercise Training Group (Experimental)
  Interventions: Other: Resistance Exercise Training Group
- Combined Exercise Training Group (Experimental)
  Interventions: Other: Combined Exercise Training Group

INTERVENTIONS:
Other: Aerobic exercise training Group — Aerobic Exercise includes Treadmill walking At Week 1-2, intensity of 40-45% Heart rate maximum (HR max), 3 days/week, for 30 minutes At Week 3-4, intensity of 45-50% HR max, 3 days /week, for 30 minutes At Week 5-6, intensity of 50-60% HR max 3 days per week, for 30 minutes
  Arms: Aerobic exercise training Group
Other: Resistance Exercise Training Group — Resistive Exercises includes (a) Leg press b) Quadriceps extension c) Bicep curl d) Hip abduction.
  At Week 1-2, 10 repetitions 1 set, 3 days/week, for 30 minutes At Week 3-4, 2 sets of 10 repetitions, 3 times /week for 30 minutes At week 5-6, 2 sets of 10 repetitions with 5 sec hold 3 times per week for 30 minutes
  Arms: Resistance Exercise Training Group
Other: Combined Exercise Training Group — Combined Exercise training includes [Aerobic: Treadmill walking + Resistive Training: a) Leg press b) Quadriceps extension c) Bicep curl d) Hip abduction] Time will be reduced to 15 minutes for both trainings in respective weeks. Aerobic Exercise includes Treadmill walking At Week 1-2, intensity of 40-45% Heart rate maximum (HR max), 3 days/week, for 15 minutes At Week 3-4, intensity of 45-50% HR max, 3 days /week, for 15 minutes At Week 5-6, intensity of 50-60% HR max 3 days per week, for 15 minutes
  Resistive Exercises At Week 1-2, 10 repetitions 1 set, 3 days/week, for 15 minutes At Week 3-4, 2 sets of 10 repetitions, 3 times /week for 15 minutes At week 5-6, 2 sets of 10 repetitions with 5 sec hold 3 times per week for 15 minutes
  Arms: Combined Exercise Training Group

SUMMARY:
To compare the effects of aerobic, resistance and combined training in hypertensive obese patients

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive with BP greater than 140/90 mmHg
* Overweight and obese adults with BMI (25-40)
* Physically inactive from past 6 months assessed with pedometer. Those with step count of less than 7000 will be included
* To be able to exercise (6MWT),t hose who completed the test without any symptom

Exclusion Criteria:

* Any active systemic illness that restricts exercise
* People doing exercise on regular basis
* Any cardiopulmonary , metabolic and neurological illness

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure | 6 weeks
  Changes from the Baseline, Blood pressure is measured through sphygmomanometer
Body Mass Index (BMI) | 6 Week
  Changes from the Baseline, Body mass index (BMI) will be calculated as weight (kg)/height (m2). Below 18.5 Underweight 18.5 - 24.9 Healthy Weight 25.0 - 29.9 Overweight 30.0 and Above Obesity
Change in blood lipid profile | 6 Week
  Change in plasma total cholesterol, high density lipoproteins cholesterol (HDL), and low density lipoproteins cholesterol (LDL) after each treatment.
Step Count | 6 week
  Pedometer is a valid self-report measure of physical activity. Pedometer is used to count the average daily steps. Change from the baseline to 6 week will be compared.
Waist circumference | 6 week
  Waist circumference will be measured for abdominal or central fat mass. It is measured in cm at the middle distance between the last floating rib and the iliac crest using a retractable ergonomic measuring tape. Change from the baseline to 6 week will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- District Headquarter Hospital - kotli, Kotli, Azad Jamu Kashmir, Pakistan

IPD SHARING:
Plan to Share IPD: No